CLINICAL TRIAL: NCT07248046
Title: Comparing Cervical Mucus, PDG, LH, and Basal Body Temperature Combinations for Ovulation and Luteal Phase Identification Using the Premom Smartphone App Versus User-Read Test Results: A Prospective Observational Study
Brief Title: Smartphone vs Manual Interpretation of Biomarkers for Ovulation and Luteal Phase Detection (SMOM Study)
Acronym: SMOM
Status: Recruiting | Type: Observational
Sponsor: Bruyère Health Research Institute. (Other)
Responsible Party: Principal Investigator, Rene Leiva, Principal Investigator, Bruyère Health Research Institute.
Other Study IDs: REB-2026-56
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Fertility; Mobile Applications; Artifical Intelligence; Cervical Mucus; Body Temperature; Luteinizing Hormone (LH); Ovulation; Menstrual Cycle; Progesterone
Keywords: Ovulation; Luteal Phase; Menstrual Cycle; Fertility; Cervical Mucus; Luteinizing Hormone; Pregnanediol Glucuronide; Progesterone; Basal Body Temperature; Female Reproductive Physiology; Fertility Awareness-Based Methods; Mobile Applications; Smartphone App; Artificial Intelligence; Self-Testing; Home Diagnostic Tests; Observational Study; Prospective Studies; Digital Health; Women's Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premom App Users: Women aged 16 to 45 already using the Premom App, who will track daily fertility signs over 3 menstrual cycles.
  Interventions: Other: Premom App-Assisted Fertility Tracking

INTERVENTIONS:
Other: Premom App-Assisted Fertility Tracking — Participants use the Premom smartphone application (Easy Healthcare Corporation) to log daily fertility indicators - cervical mucus (CM), urinary luteinizing hormone (LH) strips, urinary pregnanediol glucuronide (PDG) strips, and basal body temperature (BBT) - over three menstrual cycles. Both participant-read and AI-interpreted app readings are compared to identify ovulation and luteal phase length. **This is an observational study. Participants are not assigned to any intervention; all fertility signs collected are part of their existing self-tracking using the Premom App. The study analyzes these naturally occurring data to compare marker pairings for identifying ovulation and luteal phase length.**

SUMMARY:
This study will compare different combinations of fertility signs (cervical mucus (CM), luteinizing hormone [LH], pregnanediol glucuronide [PDG], and basal body temperature [BBT]) to determine which are most reliable for identifying ovulation and luteal phase length. Thirty existing Premom App users will track daily observations for three menstrual cycles. Participants will record mucus, perform urine tests, upload test strip photos to the Premom App, and measure BBT. Both participant readings and AI-assisted app readings will be analyzed. The main goal is to find which marker pairings give the most accurate picture of ovulation timing and luteal phase length. Secondary goals include understanding ease of use, the number of tests required, and whether the app improves accuracy.

DETAILED DESCRIPTION:
This study examines how well different combinations of fertility signs-cervical mucus changes, hormone levels in urine, and body temperature-can help identify ovulation and luteal phase length. The study uses the Premom App, which allows users to record fertility signs and take photos of urine hormone test strips for AI-assisted interpretation. Four marker pairs will be compared: Mucus plus PDG, LH plus PDG, Mucus plus BBT, and LH plus BBT. Each participant will track three cycles, with both app-based and user-based readings analyzed. The study will assess which marker pairings are most accurate and user-friendly. Secondary endpoints include usability, test burden, and app vs. participant agreement. Results may support improvements in fertility awareness and digital health tools. Risks are minimal and involve time commitment for daily tracking. **This is an observational study. Participants are not assigned to any intervention; all fertility signs collected are part of their existing self-tracking using the Premom App. The study analyzes these naturally occurring data to compare marker pairings for identifying ovulation and luteal phase length.**

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 16 to 45
* Natural menstrual cycles equal or less than 35 days
* Off hormonal contraception for more than 3 months
* Current user of the Premom App
* Willing to track cervical mucus, LH, PDG, and BBT for 3 full cycles
* Lives within 50 km of study site in the Ottawa region
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Current hormonal therapy or contraception
* Known anovulatory disorders, e.g., Polycystic Ovary Syndrome, hypothalamic amenorrhea.
* Very irregular or absent cycles
* Not using the Premom App
* Unable or unwilling to complete tracking or provide consent

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will include up to 30 adult women aged 16 to 45 years who have natural menstrual cycles and are current users of the Premom smartphone application for fertility tracking. All participants will reside within approximately 50 kilometers of Ottawa, Ontario, Canada. Participants must be off hormonal contraception for at least three months and willing to record daily fertility signs-cervical mucus, urinary LH and PDG test results, and basal body temperature-over three consecutive menstrual cycles. The study population represents healthy women of reproductive age who are already engaged in self-tracking of fertility and menstrual health using mobile technology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Agreement Between Marker Combinations and the Estimated Day of Ovulation (EDO) | Through completion of each menstrual cycle (cycle length up to 35 days), over 3 consecutive cycles per participant
  This outcome evaluates how four fertility marker combinations identify the Estimated Day of Ovulation (EDO) across three menstrual cycles. Participants will record daily cervical mucus (CM) observations, urinary luteinizing hormone (LH) and pregnanediol glucuronide (PDG) results, and basal body temperature (BBT), using both manual readings and the Premom smartphone app. For each cycle, the EDO will be established using validated physiologic indicators, including peak-type cervical mucus, the LH surge, the rise in PDG, and the post-ovulatory BBT shift. The EDO identified by each marker combination-cervical mucus plus PDG, LH plus PDG, cervical mucus plus BBT, and LH plus BBT. Agreement will be assessed by calculating the absolute day-difference between estimates.
Luteal Phase Length Determined by Different Fertility Marker Combinations | Daily tracking through completion of each menstrual cycle (cycle length up to 35 days), over 3 consecutive cycles per participant.
  Number of days from the estimated day of ovulation to the onset of the next menstrual period, calculated for each marker combination and compared within subjects across three menstrual cycles.

SECONDARY OUTCOMES:
User Satisfaction with Fertility Tracking Methods | At completion of Cycle 3 (cycle length up to 35 days).
  Participant satisfaction will be measured using the nineteen-item Participant Evaluation Survey, which examines clarity of instructions, ease of daily tracking, use of cervical mucus observations, LH and PDG tests, BBT measurements, app-based interpretation, time burden, and overall value. Each item uses a five-option Likert scale: Strongly Agree, Agree, Neutral, Disagree, and Strongly Disagree. Higher-rated responses indicate better usability, clearer instructions, lower perceived burden, and greater overall satisfaction.
Agreement Between Participant and App Interpretations of LH and PDG Test Strips | At completion of Cycle 3 (cycle length up to 35 days).
  Concordance rate between participant visual interpretation and Premom App AI-assisted interpretation of LH and PDG test strip results, expressed as percent agreement.
Testing Burden and Number of Testing Days per Cycle | Daily tracking Through completion of each menstrual cycle (cycle length up to 35 days), over 3 consecutive cycles per participant.
  Average number of days participants perform LH and PDG testing per cycle across three cycles, recorded in the study tracking log and used to evaluate practicality of each marker combination.
App Usability and Functionality Evaluation | At completion of Cycle 3 (cycle length up to 35 days).
  Participant feedback on functionality, photo upload reliability, and AI test interpretation accuracy of the Premom App, rated through the end-of-study usability survey.
Correlation Between Cervical Mucus-Defined and Standard Fertile Window | Through completion of each menstrual cycle (cycle length up to 35 days), over 3 consecutive cycles per participant.
  Comparison between fertile days identified by cervical mucus observations and the classic Wilcox fertile window (the 5 days before and including ovulation), expressed as percent overlap and mean day difference.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Laurent Ideal Clinic, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Youngster M, Luz A, Baum M, Hourvitz R, Reuvenny S, Maman E, Hourvitz A. Artificial intelligence in the service of intrauterine insemination and timed intercourse in spontaneous cycles. Fertil Steril. 2023 Nov;120(5):1004-1012. doi: 10.1016/j.fertnstert.2023.07.008. Epub 2023 Jul 23. PMID 37490977
- [Background] • Wang L, He L, Li J, Zeng D, Wen Y. T Line and C Line Detection and Ratio Reading of the Ovulation Test Strip Based on Deep Learning. In: Intelligent Data Engineering and Automated Learning - IDEAL 2021. Springer, Cham. Lecture Notes in Computer Science. 2021 Nov 23;(13113):625-636. https://www.researchgate.net/publication/356488630_T_Line_and_C_Line_Detection_and_Ratio_Reading_of_the_Ovulation_Test_Strip_Based_on_Deep_Learning
- [Background] Potluri V, Kathiresan PS, Kandula H, Thirumalaraju P, Kanakasabapathy MK, Kota Sai Pavan S, Yarravarapu D, Soundararajan A, Baskar K, Gupta R, Gudipati N, C Petrozza J, Shafiee H. An inexpensive smartphone-based device for point-of-care ovulation testing. Lab Chip. 2018 Dec 18;19(1):59-67. doi: 10.1039/c8lc00792f. PMID 30534677
- [Background] Pattnaik S, Das D, Venkatesan VA. Validation of urinary reproductive hormone measurements using a novel smartphone connected reader. Sci Rep. 2023 Jun 7;13(1):9227. doi: 10.1038/s41598-023-36539-w. PMID 37286704
- [Background] Mendizabal-Ruiz G, Paredes O, Alvarez A, Acosta-Gomez F, Hernandez-Morales E, Gonzalez-Sandoval J, Mendez-Zavala C, Borrayo E, Chavez-Badiola A. Artificial Intelligence in Human Reproduction. Arch Med Res. 2024 Dec;55(8):103131. doi: 10.1016/j.arcmed.2024.103131. Epub 2024 Nov 29. PMID 39615376
- [Background] Leiva RA, Bouchard TP, Abdullah SH, Ecochard R. Urinary Luteinizing Hormone Tests: Which Concentration Threshold Best Predicts Ovulation? Front Public Health. 2017 Nov 28;5:320. doi: 10.3389/fpubh.2017.00320. eCollection 2017. PMID 29234665
- [Background] Leiva R, Ecochard R. Helping Patients to Predict and Confirm Ovulation with the Use of Combined Urinary Hormonal and Smartphone Technology: A Proof-of-Concept Retrospective Descriptive Case Series. Semin Reprod Med. 2024 Jun;42(2):90-99. doi: 10.1055/s-0044-1791702. Epub 2024 Oct 8. PMID 39379045
- [Background] Leiva R, McNamara-Kilian M, Niezgoda H, Ecochard R, Bouchard T. Pilot observational prospective cohort study on the use of a novel home-based urinary pregnanediol 3-glucuronide (PDG) test to confirm ovulation when used as adjunct to fertility awareness methods (FAMs) stage 1. BMJ Open. 2019 May 27;9(5):e028496. doi: 10.1136/bmjopen-2018-028496. PMID 31133596
- [Background] Gibbons T, Reavey J, Georgiou EX, Becker CM. Timed intercourse for couples trying to conceive. Cochrane Database Syst Rev. 2023 Sep 15;9(9):CD011345. doi: 10.1002/14651858.CD011345.pub3. PMID 37709293
- [Background] Ecochard R, Leiva R, Bouchard T, Boehringer H, Iwaz J, Plotton I. Descriptive analysis of the relationship between progesterone and basal body temperature across the menstrual cycle. Steroids. 2022 Feb;178:108964. doi: 10.1016/j.steroids.2022.108964. Epub 2022 Jan 20. PMID 35065994
- [Background] Ecochard R, Leiva R, Bouchard T, Boehringer H, Direito A, Mariani A, Fehring R. Use of urinary pregnanediol 3-glucuronide to confirm ovulation. Steroids. 2013 Oct;78(10):1035-40. doi: 10.1016/j.steroids.2013.06.006. Epub 2013 Jul 4. PMID 23831784
- [Background] Ecochard R, Duterque O, Leiva R, Bouchard T, Vigil P. Self-identification of the clinical fertile window and the ovulation period. Fertil Steril. 2015 May;103(5):1319-25.e3. doi: 10.1016/j.fertnstert.2015.01.031. Epub 2015 Feb 24. PMID 25724738
- [Background] Duane M, Stanford JB, Porucznik CA, Vigil P. Fertility Awareness-Based Methods for Women's Health and Family Planning. Front Med (Lausanne). 2022 May 24;9:858977. doi: 10.3389/fmed.2022.858977. eCollection 2022. PMID 35685421
- [Background] Bouchard TP, Fehring RJ, Schneider M. Pilot Evaluation of a New Urine Progesterone Test to Confirm Ovulation in Women Using a Fertility Monitor. Front Public Health. 2019 Jul 2;7:184. doi: 10.3389/fpubh.2019.00184. eCollection 2019. PMID 31312631
- [Background] Bouchard TP. Using Quantitative Hormonal Fertility Monitors to Evaluate the Luteal Phase: Proof of Concept Case Study. Medicina (Kaunas). 2023 Jan 10;59(1):140. doi: 10.3390/medicina59010140. PMID 36676764
- See also: • G. Maroju R, G. Choudhari S, Shaikh MK et al. Application of artificial intelligence-based strategies for promotion of family planning in India: a scoping review [version 1; peer review: awaiting peer review]. F1000Research 2023, 12:1447 — https://doi.org/10.12688/f1000research.138006.1
- See also: • Steward K, Raja A. Physiology, Ovulation And Basal Body Temperature. [Updated 2023 Jul 17]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. — https://www.ncbi.nlm.nih.gov/books/NBK546686/